CLINICAL TRIAL: NCT03196258
Title: Cognitive Behavioural Therapy to Improve Outcomes of High Risk Patients Following Internal Fixation of Extremity Fractures: A Randomized Controlled Trial (SPOC-CBT)
Brief Title: Cognitive Behavioural Therapy to Reduce Persistent Post-Surgical Pain After Fracture
Acronym: SPOC_CBT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility issues with the study treatment (in-person CBT) resulted in the study ending earlier than anticipated.
Sponsor: McMaster University (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other); Hamilton Health Sciences Corporation (Other); Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPOC-CBT-001
Record Dates: First submitted 2017-06-13; First posted 2017-06-22 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Pain, Postoperative; Fractures, Closed; Fractures, Open
Keywords: fracture; persistent pain; cognitive behavioural therapy; post surgical pain; health-related quality of life
MeSH Terms: conditions — Pain, Postoperative; Fractures, Closed; Fractures, Open; Fractures, Bone | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants with operatively managed extremity fractures who screen positive for unhelpful illness beliefs (SPOC scores ≥78) 6-weeks post-fracture fixation will be randomized to receive either 6 weekly one-on-one, 1-hour sessions of cognitive behavioral therapy (CBT) or standard of care (control). Outcomes will be assessed at 3 months, 6 months, 9 months, and 12 months' post-fracture
Masking Description: Eligible participants will be randomized to 1 of 2 groups: 1) CBT intervention or 2) standard of care. Due to the nature of the intervention, it will not be feasible to blind participants, treating surgeons, or CBT therapists to treatment allocation. The data analyst and Steering Committee will be blinded to treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention - CBT (Experimental): Participants in this arm will receive 6 weekly one-on-one, 1-hour sessions of Cognitive Behavioural Therapy session (intervention) in addition to receiving standard of care treatment for their fracture(s).
  Interventions: Behavioral: Cognitive behavioural therapy
- control (No Intervention): Participants in the control arm of the study will receive standard of care treatment for their fracture(s) but will not receive any Cognitive Behavioral Therapy.

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy — Participants who are randomized to the CBT intervention are required to start CBT within 8 weeks of their fracture surgery. The CBT intervention will consist of 6 weekly one-on-one, 1-hour sessions that will focus on addressing maladaptive beliefs related to pain and recovery as well as teaching skills to enhance coping and management of pain symptoms. The specific focus of CBT sessions will be informed by each individual patient's responses on the SPOC questionnaire. All other aspects of post-operative care will be at the discretion of participant's surgeon
  Other Names: CBT
  Arms: intervention - CBT

SUMMARY:
Psychological factors such as stress, distress, anxiety, depression, and poor coping strategies may be associated with ongoing pain following injuries such as fractures. In order to study this relationship, researchers at McMaster University have developed the Somatic Pre-Occupation and Coping (SPOC) questionnaire, which identifies illness beliefs that may help to predict which patients are at risk for ongoing pain, reduced quality of life, and delays in returning to work and leisure activities after a fracture requiring surgical treatment. Previous research using the SPOC questionnaire suggests the possibility that fracture patients with illness beliefs that put them at risk for developing ongoing pain could be identified early in the treatment process. These patients may benefit from cognitive behavioural therapy (CBT) which is designed to modify such thoughts with the goal of reducing ongoing pain and improving quality of life. The goal of this study is to determine if CBT is effective in reducing ongoing pain and improving quality of life in fracture patients who show illness beliefs that may place them at risk for developing ongoing pain.

DETAILED DESCRIPTION:
In North America, chronic non-cancer pain affects approximately 30% of the population, with similar rates in Europe and Australia. Surgery and trauma are frequently cited as triggering events responsible for the development of chronic pain. A survey of 5,130 patients attending 10 outpatient clinics located throughout North Britain found that 41% attributed their chronic pain to a traumatic event or surgery. The presence of persistent pain can have a major impact on patients' quality of life, including their ability to return to work and their daily activities.

The relationship between psychological factors, behaviors, and cognitive processes and the sensation of pain is well documented. Stress, distress, anxiety, depression, catastrophizing, fear-avoidance behaviors, and poor coping strategies appear to have a significant positive relationship with both acute and chronic pain. Evidence suggests that these psychological factors can cause alterations along the spinal and supraspinal pain pathways which influence the perception of pain. Previous studies suggest that patients' beliefs and expectations may be associated with clinical outcomes, including self-reported pain.

Clinical outcomes following operatively managed fractures of the extremities are variable and many patients continue to experience persistent pain and disability one-year after surgery and beyond. In a recent trial involving patients with open extremity fractures, 65% of patients reported moderate to very severe pain and 35% reported moderate to extreme pain interference at one-year. A systematic review of 20 observational studies of traumatic tibial fracture repairs found the mean incidence of persistent post-surgical pain (PPSP) was 47.4% (range: 10% to 86%) at an average of 23.9 months after surgery. Although several risk factors for PPSP have been identified, many, such as younger age and female gender, are non-modifiable and thus not amendable to direct intervention.

The effect of patients' beliefs and expectations on their recovery following traumatic injuries is an under-investigated area. In response to this gap, Busse et al. developed and evaluated the Somatic Pre-Occupation and Coping (SPOC) questionnaire to identify unhelpful illness beliefs that are predictive of poorer functional outcomes post-fracture. This self-administered questionnaire identified unhelpful illness beliefs among approximately one third of patients with operatively managed extremity fractures. Furthermore, high somatic pre-occupation and poor coping at 6-weeks post-fracture (as measured by the SPOC questionnaire) were found to be strongly associated with PPSP, functional limitations, unemployment, and reduced quality of life 1 year after fracture fixation. This suggests the possibility that fracture patients who exhibit unhelpful illness beliefs can be identified and targeted for concurrent therapy designed to modify such cognitions and improve prognosis. At present, however, there are no approaches that have been shown effective for improving recovery among high-risk patients.

The findings from the FLOW trial highlight the importance of patient beliefs in recovery from orthopaedic trauma. A number of systematic reviews have shown patients' perceptions regarding their illness experience can be modified, and that such efforts can improve outcomes. Moss-Morris and colleagues explored the effect of CBT among patients attending a multidisciplinary chronic pain clinic and found that changes in cognitive processes accounted for 26% of the variation in improved health-related quality of life scores. Collectively, these findings suggest that targeting and modifying unhelpful beliefs through CBT may provide an effective strategy to improve outcomes among high-risk trauma patients.

ELIGIBILITY:
The inclusion criteria are:

1. Adult men or women aged 18 years and older.
2. Acute open or closed fracture(s) of the appendicular skeleton. Patients with multiple fractures may be included.
3. Fracture treated operatively with internal fixation.
4. Screened for eligibility within 6 weeks of their fracture.
5. Cognitive ability and language skills required to participate in the CBT intervention (in the judgement of site research personnel).
6. Able to start the CBT within 8 weeks of their fracture surgery.
7. Provision of informed consent.
8. Screen positive for unhelpful illness beliefs (SPOC scores ≥74), as assessed at 6 weeks' post-surgical fixation.

The exclusion criteria are:

1. Fragility fracture.
2. Stress fracture.
3. Concomitant injury which, in the opinion of the attending surgeon, is likely to impair function for as long as or longer than the patient's extremity fracture.
4. Active psychosis.
5. Active suicidality.
6. Active substance use disorder that, in the judgement of the treating surgeon, would interfere in the patient's ability to partake in the CBT and/or the study.
7. Already participating in, or planning to start other psychological treatments (including CBT) within the duration of the study (12 months).
8. Anticipated problems with the patient attending CBT sessions and/or returning for follow-up.
9. Incarceration.
10. Other reason to exclude the patient, as specified.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of Persistent Post-Surgical Pain at 12 months' post-fracture | 12 months post-fracture
  The primary outcomes are 1) PPSP according to the World Health Organization's (WHO) proposed definition, and 2) the prevalence of moderate to severe pain interference over 12 months post-fracture as assessed by an individual item from the Patient-Reported Outcomes Measurement Information System (PROMIS).
  The WHO's definition requires 4 criteria for the diagnosis of PPSP: 1) Pain that began after surgery or a tissue trauma is experienced; 2) The pain is in an area of preceding surgery or tissue trauma, 3) The pain persisted for at least two months after the initiating event, and 4) The pain is not better explained by an infection, a malignancy, a pre-existing pain condition or any other alternative cause.

SECONDARY OUTCOMES:
Short Form 12 (SF-12) | 1 year
  General health related quality of life will be assessed by the SF-12. The SF-12 is an established, reliable and validated health status measure.It is a self-administered, 12-item questionnaire that measures health-related quality of life in 8 domains related to physical, social, mental, and emotional functioning, bodily pain, and general health. Both physical and mental summary scores can be obtained. Each domain is scored separately from 0 (lowest level) to 100 (highest level).
Return to Function questionnaire | 1 year
  Return to function will be measured by when participants' return to work, household activities, and leisure activities, as well as when they achieve 80% of their pre-injury function. The return to function outcome will be assessed using the Return to Function questionnaire.
PROMIS-Physical Function 28 | 1 year
  HRQL will also be assessed by the PROMIS-PF28, as recent research suggests it may be more sensitive to change than the SF-12. The PROMIS-PF is a standard for patient-reported outcomes research and practice and recommended for initial outcome assessment. Studies continue to support its construct validity and feasibility. The PROMIS-PF includes seven HRQoL domains: Physical Functioning, Anxiety, Depression, Fatigue, Sleep Disturbance, Social Functioning, and Pain. The PROMIS-Physical Function 28 will be used to assess seven health quality of life domains.

OTHER OUTCOMES:
Exploratory outcome 1: Fracture healing complications | 1 year
  fracture healing complications as assessed by the treating surgeon (including wound healing problems, infection (superficial and deep), hardware failure, hardware breakage, and non-union),
Exploratory outcome 2: time to fracture healing | 1 year
  time to clinical fracture healing, as assessed by the treating surgeon. To determine if CBT versus usual care reduces the incidence of fracture healing complications within 12-months post-fracture
Exploratory outcome 3: opioid use | 1 year
  Patient-reported use of opioid class medications. ) to determine if CBT versus usual care reduces the proportion of participants taking opioid class medications at 6 months and 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moulin DE, Clark AJ, Speechley M, Morley-Forster PK. Chronic pain in Canada--prevalence, treatment, impact and the role of opioid analgesia. Pain Res Manag. 2002 Winter;7(4):179-84. doi: 10.1155/2002/323085. PMID 12518174
- [Background] Johannes CB, Le TK, Zhou X, Johnston JA, Dworkin RH. The prevalence of chronic pain in United States adults: results of an Internet-based survey. J Pain. 2010 Nov;11(11):1230-9. doi: 10.1016/j.jpain.2010.07.002. Epub 2010 Aug 25. PMID 20797916
- [Background] Blyth FM, March LM, Brnabic AJ, Jorm LR, Williamson M, Cousins MJ. Chronic pain in Australia: a prevalence study. Pain. 2001 Jan;89(2-3):127-34. doi: 10.1016/s0304-3959(00)00355-9. PMID 11166468
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934
- [Background] Elliott AM, Smith BH, Penny KI, Smith WC, Chambers WA. The epidemiology of chronic pain in the community. Lancet. 1999 Oct 9;354(9186):1248-52. doi: 10.1016/s0140-6736(99)03057-3. PMID 10520633
- [Background] Crombie IK, Davies HT, Macrae WA. Cut and thrust: antecedent surgery and trauma among patients attending a chronic pain clinic. Pain. 1998 May;76(1-2):167-71. PMID 9696470
- [Background] Linton SJ. A review of psychological risk factors in back and neck pain. Spine (Phila Pa 1976). 2000 May 1;25(9):1148-56. doi: 10.1097/00007632-200005010-00017. PMID 10788861
- [Background] Wiech K, Tracey I. The influence of negative emotions on pain: behavioral effects and neural mechanisms. Neuroimage. 2009 Sep;47(3):987-94. doi: 10.1016/j.neuroimage.2009.05.059. Epub 2009 May 28. PMID 19481610
- [Background] Mondloch MV, Cole DC, Frank JW. Does how you do depend on how you think you'll do? A systematic review of the evidence for a relation between patients' recovery expectations and health outcomes. CMAJ. 2001 Jul 24;165(2):174-9. PMID 11501456
- [Background] Ebrahim S, Malachowski C, Kamal El Din M, Mulla SM, Montoya L, Bance S, Busse JW. Measures of patients' expectations about recovery: a systematic review. J Occup Rehabil. 2015 Mar;25(1):240-55. doi: 10.1007/s10926-014-9535-4. PMID 25100443
- [Background] Sprague S, Leece P, Bhandari M, Tornetta P 3rd, Schemitsch E, Swiontkowski MF; S.P.R.I.N.T. Investigators. Limiting loss to follow-up in a multicenter randomized trial in orthopedic surgery. Control Clin Trials. 2003 Dec;24(6):719-25. doi: 10.1016/j.cct.2003.08.012. PMID 14662277
- [Background] Montes A, Roca G, Sabate S, Lao JI, Navarro A, Cantillo J, Canet J; GENDOLCAT Study Group. Genetic and Clinical Factors Associated with Chronic Postsurgical Pain after Hernia Repair, Hysterectomy, and Thoracotomy: A Two-year Multicenter Cohort Study. Anesthesiology. 2015 May;122(5):1123-41. doi: 10.1097/ALN.0000000000000611. PMID 25985024
- [Background] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770
- [Background] Busse JW, Bhandari M, Guyatt GH, Heels-Ansdell D, Kulkarni AV, Mandel S, Sanders D, Schemitsch E, Swiontkowski M, Tornetta P 3rd, Wai E, Walter SD; SPRINT Investigators & the Medically Unexplained Syndromes Study Group. Development and validation of an instrument to predict functional recovery in tibial fracture patients: the Somatic Pre-Occupation and Coping (SPOC) questionnaire. J Orthop Trauma. 2012 Jun;26(6):370-8. doi: 10.1097/BOT.0b013e31822421e2. PMID 22011635
- [Background] Reininga IH, Brouwer S, Dijkstra A, Busse JW, Ebrahim S, Wendt KW, El Moumni M. Measuring illness beliefs in patients with lower extremity injuries: reliability and validity of the Dutch version of the Somatic Pre-Occupation and Coping questionnaire (SPOC-NL). Injury. 2015 Feb;46(2):308-14. doi: 10.1016/j.injury.2014.08.042. Epub 2014 Sep 16. PMID 25441575
- [Background] Bhandari M, Petrisor BA, Jeray KJ. Wound Irrigation in Initial Management of Open Fractures. N Engl J Med. 2016 May 5;374(18):1789-90. doi: 10.1056/NEJMc1601157. No abstract available. PMID 27144859
- [Background] Brodke DJ, Saltzman CL, Brodke DS. PROMIS for Orthopaedic Outcomes Measurement. J Am Acad Orthop Surg. 2016 Nov;24(11):744-749. doi: 10.5435/JAAOS-D-15-00404. PMID 27661391
- [Background] Werner MU, Kongsgaard UE. I. Defining persistent post-surgical pain: is an update required? Br J Anaesth. 2014 Jul;113(1):1-4. doi: 10.1093/bja/aeu012. Epub 2014 Feb 18. No abstract available. PMID 24554546
- [Background] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Khan JS, Devereaux PJ, LeManach Y, Busse JW. Patient coping and expectations about recovery predict the development of chronic post-surgical pain after traumatic tibial fracture repair. Br J Anaesth. 2016 Sep;117(3):365-70. doi: 10.1093/bja/aew225. PMID 27543531
- [Background] Lin CA, Swiontkowski M, Bhandari M, Walter SD, Schemitsch EH, Sanders D, Tornetta P 3rd. Reaming Does Not Affect Functional Outcomes After Open and Closed Tibial Shaft Fractures: The Results of a Randomized Controlled Trial. J Orthop Trauma. 2016 Mar;30(3):142-8. doi: 10.1097/BOT.0000000000000497. PMID 26618662
- [Background] Katsoulis E, Court-Brown C, Giannoudis PV. Incidence and aetiology of anterior knee pain after intramedullary nailing of the femur and tibia. J Bone Joint Surg Br. 2006 May;88(5):576-80. doi: 10.1302/0301-620X.88B5.16875. No abstract available. PMID 16645100
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] MacKenzie EJ, Bosse MJ, Kellam JF, Pollak AN, Webb LX, Swiontkowski MF, Smith DG, Sanders RW, Jones AL, Starr AJ, McAndrew MP, Patterson BM, Burgess AR, Travison T, Castillo RC. Early predictors of long-term work disability after major limb trauma. J Trauma. 2006 Sep;61(3):688-94. doi: 10.1097/01.ta.0000195985.56153.68. PMID 16967009
- [Background] Wegener ST, Castillo RC, Haythornthwaite J, MacKenzie EJ, Bosse MJ; LEAP Study Group. Psychological distress mediates the effect of pain on function. Pain. 2011 Jun;152(6):1349-1357. doi: 10.1016/j.pain.2011.02.020. Epub 2011 Mar 10. PMID 21396777
- [Background] Vranceanu AM, Bachoura A, Weening A, Vrahas M, Smith RM, Ring D. Psychological factors predict disability and pain intensity after skeletal trauma. J Bone Joint Surg Am. 2014 Feb 5;96(3):e20. doi: 10.2106/JBJS.L.00479. PMID 24500592
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. A classification of chronic pain for ICD-11. Pain. 2015 Jun;156(6):1003-1007. doi: 10.1097/j.pain.0000000000000160. No abstract available. PMID 25844555
- [Background] Fries JF, Bruce B, Cella D. The promise of PROMIS: using item response theory to improve assessment of patient-reported outcomes. Clin Exp Rheumatol. 2005 Sep-Oct;23(5 Suppl 39):S53-7. PMID 16273785
- [Background] Angst F, Aeschlimann A, Stucki G. Smallest detectable and minimal clinically important differences of rehabilitation intervention with their implications for required sample sizes using WOMAC and SF-36 quality of life measurement instruments in patients with osteoarthritis of the lower extremities. Arthritis Rheum. 2001 Aug;45(4):384-91. doi: 10.1002/1529-0131(200108)45:43.0.CO;2-0. PMID 11501727
- [Background] Jenkinson C, Stewart-Brown S, Petersen S, Paice C. Assessment of the SF-36 version 2 in the United Kingdom. J Epidemiol Community Health. 1999 Jan;53(1):46-50. doi: 10.1136/jech.53.1.46. PMID 10326053
- [Background] Fixation using Alternative Implants for the Treatment of Hip fractures (FAITH) Investigators. Fracture fixation in the operative management of hip fractures (FAITH): an international, multicentre, randomised controlled trial. Lancet. 2017 Apr 15;389(10078):1519-1527. doi: 10.1016/S0140-6736(17)30066-1. Epub 2017 Mar 3. PMID 28262269
- [Background] Madden K, Scott T, McKay P, Petrisor BA, Jeray KJ, Tanner SL, Bhandari M, Sprague S. Predicting and Preventing Loss to Follow-up of Adult Trauma Patients in Randomized Controlled Trials: An Example from the FLOW Trial. J Bone Joint Surg Am. 2017 Jul 5;99(13):1086-1092. doi: 10.2106/JBJS.16.00900. PMID 28678121
- [Background] Zhang Y, Alyass A, Vanniyasingam T, Sadeghirad B, Florez ID, Pichika SC, Kennedy SA, Abdulkarimova U, Zhang Y, Iljon T, Morgano GP, Colunga Lozano LE, Aloweni FAB, Lopes LC, Yepes-Nunez JJ, Fei Y, Wang L, Kahale LA, Meyre D, Akl EA, Thabane L, Guyatt GH. A systematic survey of the methods literature on the reporting quality and optimal methods of handling participants with missing outcome data for continuous outcomes in randomized controlled trials. J Clin Epidemiol. 2017 Aug;88:67-80. doi: 10.1016/j.jclinepi.2017.05.016. Epub 2017 Jun 1. PMID 28579378
- [Background] Thabane L, Mbuagbaw L, Zhang S, Samaan Z, Marcucci M, Ye C, Thabane M, Giangregorio L, Dennis B, Kosa D, Borg Debono V, Dillenburg R, Fruci V, Bawor M, Lee J, Wells G, Goldsmith CH. A tutorial on sensitivity analyses in clinical trials: the what, why, when and how. BMC Med Res Methodol. 2013 Jul 16;13:92. doi: 10.1186/1471-2288-13-92. PMID 23855337
- [Background] Sprague S, Petrisor BA, Jeray KJ, McKay P, Scott T, Heels-Ansdell D, Schemitsch EH, Liew S, Guyatt GH, Walter SD, Bhandari M. Factors Associated With Health-Related Quality of Life in Patients With Open Fractures. J Orthop Trauma. 2018 Jan;32(1):e5-e11. doi: 10.1097/BOT.0000000000000993. PMID 28799963
- [Background] Archer KR, Abraham CM, Obremskey WT. Psychosocial Factors Predict Pain and Physical Health After Lower Extremity Trauma. Clin Orthop Relat Res. 2015 Nov;473(11):3519-26. doi: 10.1007/s11999-015-4504-6. PMID 26282387
- [Background] Sun X, Briel M, Walter SD, Guyatt GH. Is a subgroup effect believable? Updating criteria to evaluate the credibility of subgroup analyses. BMJ. 2010 Mar 30;340:c117. doi: 10.1136/bmj.c117. No abstract available. PMID 20354011
- [Background] Briggs AH, O'Brien BJ, Blackhouse G. Thinking outside the box: recent advances in the analysis and presentation of uncertainty in cost-effectiveness studies. Annu Rev Public Health. 2002;23:377-401. doi: 10.1146/annurev.publhealth.23.100901.140534. Epub 2001 Oct 25. PMID 11910068
- [Background] Briel M, Lane M, Montori VM, Bassler D, Glasziou P, Malaga G, Akl EA, Ferreira-Gonzalez I, Alonso-Coello P, Urrutia G, Kunz R, Culebro CR, da Silva SA, Flynn DN, Elamin MB, Strahm B, Murad MH, Djulbegovic B, Adhikari NK, Mills EJ, Gwadry-Sridhar F, Kirpalani H, Soares HP, Abu Elnour NO, You JJ, Karanicolas PJ, Bucher HC, Lampropulos JF, Nordmann AJ, Burns KE, Mulla SM, Raatz H, Sood A, Kaur J, Bankhead CR, Mullan RJ, Nerenberg KA, Vandvik PO, Coto-Yglesias F, Schunemann H, Tuche F, Chrispim PP, Cook DJ, Lutz K, Ribic CM, Vale N, Erwin PJ, Perera R, Zhou Q, Heels-Ansdell D, Ramsay T, Walter SD, Guyatt GH. Stopping randomized trials early for benefit: a protocol of the Study Of Trial Policy Of Interim Truncation-2 (STOPIT-2). Trials. 2009 Jul 6;10:49. doi: 10.1186/1745-6215-10-49. PMID 19580665
- [Background] Montori VM, Devereaux PJ, Adhikari NK, Burns KE, Eggert CH, Briel M, Lacchetti C, Leung TW, Darling E, Bryant DM, Bucher HC, Schunemann HJ, Meade MO, Cook DJ, Erwin PJ, Sood A, Sood R, Lo B, Thompson CA, Zhou Q, Mills E, Guyatt GH. Randomized trials stopped early for benefit: a systematic review. JAMA. 2005 Nov 2;294(17):2203-9. doi: 10.1001/jama.294.17.2203. PMID 16264162
- [Derived] Gouveia K, Sprague S, Gallant J, Del Fabbro G, Leonard J, Bzovsky S, McKay P, Busse JW; COPE Investigators. In-person cognitive behavioural therapy vs. usual care after surgical management of extremity fractures: an unsuccessful feasibility trial. Pilot Feasibility Stud. 2024 Jan 6;10(1):2. doi: 10.1186/s40814-023-01430-y. PMID 38184642
- See also: 28. Hamner J, Dewitt B. The Development of a Preference-based Scoring System for PROMIS (PROPr): A Technical Report v 1.1. [Internet] 2017;available from: http://janelhanmer.pitt.edu/documents/technicalreportv1.1.pdf (accessed August 29, 2017). — http://janelhanmer.pitt.edu/ProPr.html
- See also: Wang L, Chang Y, Kennedy SA, Hong PJ, Chow N, Coubon R et al. Perioperative Psychotherapy for Persistent Post-Surgical Pain and Physical Impairment: A Meta-Analysis of Randomized Trials. Br J Anaesth. 2017;[in review] — https://www.google.ca/search?q=Wang+L%2C+Chang+Y%2C+Kennedy+SA%2C+Hong+PJ%2C+Chow+N%2C+Coubon+R+et+al.+Perioperative+Psychotherapy+for+Persistent+Post-Surgical+Pain+and+Physical+Impairment%3A+A+Meta-Analysis+of+Randomized+Trials.+Br+J+Anaesth.+2017%3B%5Bin+review%5D&oq=Wang+L%2C+Chang+Y%2C+Kennedy+SA%2C+Hong+PJ%2C+Chow+N%2C+Coubon+R+et+al.+Perioperative+Psychotherapy+for+Persistent+Post-Surgical+Pain+and+Physical+Impairment%3A+A+Meta-Analysis+of+Randomized+Trials.+Br+J+Anaesth.+2017%3B%5Bin+review%5D&aqs=chrome..69i57.453j0j9&sourceid=chrome&ie=UTF-8
- See also: Hamner J, Dewitt B. The Development of a Preference-based Scoring System for PROMIS (PROPr): A Technical Report v 1.1 [internet] 2017; available from: http//janelhanmer.pitt.edu/documents/technicalreportv1.1.pdf (accessed August 29, 2017) — http://janelhanmer.pitt.edu/ProPr.html
- See also: 33. Busse JW, Bhandari M, Einhorn TA, Schemitsch E, Heckman JD, Tornetta P, 3rd, et al. Re-evaluation of low intensity pulsed ultrasound in treatment of tibial fractures (TRUST): randomized clinical trial. Bmj. 2016;355:i5351 — http://www.bmj.com/content/355/bmj.i5351